CLINICAL TRIAL: NCT02539836
Title: Study on Dietary Nutrition Intervention Techniques for Children Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Shenzhen Children's Hospital (Other Government)
Responsible Party: Principal Investigator, Yonglong Pan, Research associate, Chinese Academy of Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: COIF_001
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Obesity; Intestinal Bacteria Flora Disturbance; Body Weight
Keywords: children's obesity; gut microbiome; body mass index; fruit and vegetable fermentation extraction; dietary nutrition intervention
MeSH Terms: conditions — Obesity; Body Weight | interventions — Magnetic Resonance Imaging; Positron-Emission Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Obesity with dietary nutrition (Experimental): Obese children will be intervented by dietary nutrition based on plant fermentation extract for 2 months.
  Interventions: Dietary Supplement: Dietary nutrition based on plant fermentation extract
- Liver fat of obese children (Active Comparator): To investigate the accuracy of MRI in quantifying liver fat with magnetic resonance spectroscopy (MRS) as a reference.
  Interventions: Diagnostic Test: MRI in quantifying liver fat with MRS

INTERVENTIONS:
Dietary Supplement: Dietary nutrition based on plant fermentation extract — The main ingredient of dietary nutrition is plant fermentation extraction which is from many fruit and vegetable fermented by probiotics.
  Arms: Obesity with dietary nutrition
Diagnostic Test: MRI in quantifying liver fat with MRS — To investigate the accuracy of MRI in quantifying liver fat with magnetic resonance spectroscopy (MRS) as a reference.
  Arms: Liver fat of obese children

SUMMARY:
With the rapid development of society and economy, children's simple obesity is the rising in the world and has become a chronic disease which is one of the biggest public health challenges in the world. It is a serious threat to the health of children and their adulthood. The overweight and obesity is induced by the genetic and environmental factors. The environmental factors are very important, while the dietary factors are the driving factors of many chronic diseases including obesity. This study focus on the dietary intervention of childhood obesity to build healthy intestinal flora. The interventing food was based on a natural health food - fruit and vegetable fermentation liquid, and combined with other probiotic dietary factors, dietary fiber and oligosaccharides. The implementation of the study will help to reveal the fuction mechanism of intestinal bacteria in the obese children and normal children, and to construct healthy micro environment of intestinal flor. According to the positive effect factors, the study will propose a healthy diet and nutrition intervention model for obese children, which is significant to social health especially to children's health.

To investigate the accuracy of MRI in quantifying liver fat with magnetic resonance spectroscopy (MRS) as a reference. A secondary goal was to assess the prevalence of nonalcoholic fatty liver disease in overweight and obese Chinese children and adolescents.

DETAILED DESCRIPTION:
Before academic examination, letter to parents, informed consent and volunteer questionnaire are released to school children and their guardians. We tell the volunteers and their guardians what about this study and invite them to participate this study. Only the volunteers and guardians signature on the letter to parents and informed consent are able to the research objects.

Experimental procedures:

Two times of medical exams, blood and stool sample collection is required for the whole experiment research. The first time exams and sample collection is carried on during academic examination; the second time is carried on after the intervention.

Recruit of research objects:

According to academic examination and volunteer questionnaires, about 300 healthy children without in taking antibiotics before 3 months are recruited and their BMI should be in the obese range. Then their waist circumference and the ratio of body fat are measured. If the ratio of waist size to weight of them is >0.46 and they have higher percentage of body fat (>20% for boys and under 12 years old girls, >25% for 12 years old girls), the data are collected and input to the database. About 40 healthy children between 15-18 years old are recruited to participate the next intervention research.

General body examination:

In academic examination, the student's basic medical data including height and weight are recorded, and then their BMI are calculated. If his/her BMI are in the obese range, his/her body composition are measured and recorded.

MRI and MRS test:

All patients underwent MRI scanning performed by an experienced technologist using a 3 Tesla MR unit (MAGNETOM Skyra, Siemens Healthcare, Erlangen, Germany). MRI and MRS were performed with multi-echo Dixon and HISTO sequences, respectively, to calculate hepatic proton density fat fraction (PDFF).

Blood collection, preservation and test:

Blood collection and preservation are proceed in standard of medical examination. When collecting the data of obesity, the tests of blood count, blood glucose, serum lipid and liver function should be processed for obese children. When intervening, more tests including blood count, blood glucose, blood lipids, liver function, hemoglobin, cytokines, insulin, high sensitivity C-reactive protein, leptin and somatomedin C should be processed.

Stool collection, preservation and detection:

50 ml centrifuge tubes are used to collect stool samples. Each tube is marked a unique encoding corresponds to a volunteer. When volunteers collecting stool samples, they transfer the stool samples into sterile centrifuge tube using sterile swabs or toothpicks as soon as possible. The collecting samples should be more than 10g. The centrifuge tubes should be put in low-temperature place , then transfer to refrigerator and stored at -80 ℃ until to DNA extraction and other testing. The tests including short chain fatty acids content (SCFA), pH, water content, immune factors sIgA and Calprotectin are processed.

16S rRNA gene sequencing of bacteria in stools:

DNA extraction:

For each sample, about 0.2g stool is weighted and the total DNA is extracted using fecal genomic DNA extraction Kit (Qiagen, model DP328). And then the concentration and purity of extracted DNA were measured using NanoDrop (Thermo, 2000C) to guarantee each sample meets the sequencing requirement.

Sample sequencing:

PCR amplification of 16S rRNA gene (V3-V4) are performed with universal forward primers 5'-ACTCCTACGGGAGGCAGCAG-3' and reverse primer 5'-GGACTACVSGGGTATCTAAT-3'. The amplification system include sterile water 19.375 ul, buffer 2.5ul, template 1ul, primers 1ul, Pyrobest DNA polymerase 0.125ul. PCR cycling conditions were as follows: 94 ℃ 5min, followed by some cycles including 94℃ denaturing for 30s, 50℃ renaturing for 30s,72℃ extending for 30s, then 72℃ extending for 5min. PCR product electrophoresis are performed to determine the appropriate PCR product with different application cycles. After connecting amplified products to tagged primers and labels, paired-end sequencing are performed with the sequencing platform of Illumina MiSeq, and the read length is about 250bp.

Intervention treatment on childhood obesity with PFE:

After 16S rRNA gene sequencing, about 40 obese volunteers in high school and with similar intestinal flora profiles are selected to participate the intervention treatment research. The intervening food is "Dr. Ephraim" plant fermentation extract (PFE). Without changing the previous diets of research objects, each research object drinks drinking 30mL PFE at morning and evening enzymes respectively, and the intervention last for 8 weeks. Before and after 8-week intervention, stool and blood samples of research objects are collected and analyzed to obtain their physiological and biochemical indexes. The all 16S rRNA gene of fecal samples in each stage are sequenced.

ELIGIBILITY:
Inclusion Criteria:

* People whose BMI>27 and Age between 15-18;the value of waistline/weight >0.46; the value of body composition >20%.

Exclusion Criteria:

* People treated by antibiotic drugs in 3 months;People with gastrointestinal diseases;People with Type I diabetes, any eating disorders such as bulimia or anorexia nervosa; Prader-Willi patients and obesity is part of clinical syndrome with other disorders.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2015-09-01; Primary Completion 2016-12-30 (Actual); Study Completion 2018-07-20 (Actual)

PRIMARY OUTCOMES:
BMI change | 2 months

SECONDARY OUTCOMES:
Serum biomarkers change | 2 months
Weight loss | 2 months
Gut microbiome profile change | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liang, Ph.D, Study Director — Shenzhen Institutes of Advanced Technology
Locations (1):
- Shenzhen Meilin High School, Shenzhen, Guangdong, China

REFERENCES:
- [Background] Tsiros MD, Coates AM, Howe PR, Grimshaw PN, Buckley JD. Obesity: the new childhood disability? Obes Rev. 2011 Jan;12(1):26-36. doi: 10.1111/j.1467-789X.2009.00706.x. PMID 20070542
- [Background] Brien SE, Katzmarzyk PT. Physical activity and the metabolic syndrome in Canada. Appl Physiol Nutr Metab. 2006 Feb;31(1):40-7. doi: 10.1139/h05-024. PMID 16604140
- [Background] Heitmann BL, Koplan J, Lissner L. Childhood obesity: successes and failures of preventive interventions. Nutr Rev. 2009 May;67 Suppl 1:S89-93. doi: 10.1111/j.1753-4887.2009.00167.x. PMID 19453687
- [Background] Aranceta J, Moreno B, Moya M, Anadon A. Prevention of overweight and obesity from a public health perspective. Nutr Rev. 2009 May;67 Suppl 1:S83-8. doi: 10.1111/j.1753-4887.2009.00166.x. PMID 19453686
- [Background] Ezzati M, Lopez AD, Rodgers A, Vander Hoorn S, Murray CJ; Comparative Risk Assessment Collaborating Group. Selected major risk factors and global and regional burden of disease. Lancet. 2002 Nov 2;360(9343):1347-60. doi: 10.1016/S0140-6736(02)11403-6. PMID 12423980
- [Background] Xu H, Li Y, Liu A, Zhang Q, Hu X, Fang H, Li T, Guo H, Li Y, Xu G, Ma J, Du L, Ma G. Prevalence of the metabolic syndrome among children from six cities of China. BMC Public Health. 2012 Jan 6;12:13. doi: 10.1186/1471-2458-12-13. PMID 22225617
- [Background] Whitaker RC, Wright JA, Pepe MS, Seidel KD, Dietz WH. Predicting obesity in young adulthood from childhood and parental obesity. N Engl J Med. 1997 Sep 25;337(13):869-73. doi: 10.1056/NEJM199709253371301. PMID 9302300
- [Background] Musso G, Gambino R, Cassader M. Obesity, diabetes, and gut microbiota: the hygiene hypothesis expanded? Diabetes Care. 2010 Oct;33(10):2277-84. doi: 10.2337/dc10-0556. PMID 20876708
- [Background] Smith JD, Montano Z, Dishion TJ, Shaw DS, Wilson MN. Preventing weight gain and obesity: indirect effects of the family check-up in early childhood. Prev Sci. 2015 Apr;16(3):408-19. doi: 10.1007/s11121-014-0505-z. PMID 25263212
- [Background] Chaput JP, Despres JP, Bouchard C, Tremblay A. Longer sleep duration associates with lower adiposity gain in adult short sleepers. Int J Obes (Lond). 2012 May;36(5):752-6. doi: 10.1038/ijo.2011.110. Epub 2011 Jun 7. PMID 21654631
- [Background] Zemel MB, Thompson W, Milstead A, Morris K, Campbell P. Calcium and dairy acceleration of weight and fat loss during energy restriction in obese adults. Obes Res. 2004 Apr;12(4):582-90. doi: 10.1038/oby.2004.67. PMID 15090625
- [Background] Chaput JP, Leblanc C, Perusse L, Despres JP, Bouchard C, Tremblay A. Risk factors for adult overweight and obesity in the Quebec Family Study: have we been barking up the wrong tree? Obesity (Silver Spring). 2009 Oct;17(10):1964-70. doi: 10.1038/oby.2009.116. Epub 2009 Apr 9. PMID 19360005
- [Background] Bervoets L, Van Hoorenbeeck K, Kortleven I, Van Noten C, Hens N, Vael C, Goossens H, Desager KN, Vankerckhoven V. Differences in gut microbiota composition between obese and lean children: a cross-sectional study. Gut Pathog. 2013 Apr 30;5(1):10. doi: 10.1186/1757-4749-5-10. PMID 23631345
- [Background] Backhed F, Ding H, Wang T, Hooper LV, Koh GY, Nagy A, Semenkovich CF, Gordon JI. The gut microbiota as an environmental factor that regulates fat storage. Proc Natl Acad Sci U S A. 2004 Nov 2;101(44):15718-23. doi: 10.1073/pnas.0407076101. Epub 2004 Oct 25. PMID 15505215
- [Background] Backhed F, Manchester JK, Semenkovich CF, Gordon JI. Mechanisms underlying the resistance to diet-induced obesity in germ-free mice. Proc Natl Acad Sci U S A. 2007 Jan 16;104(3):979-84. doi: 10.1073/pnas.0605374104. Epub 2007 Jan 8. PMID 17210919
- [Background] Turnbaugh PJ, Gordon JI. The core gut microbiome, energy balance and obesity. J Physiol. 2009 Sep 1;587(Pt 17):4153-8. doi: 10.1113/jphysiol.2009.174136. Epub 2009 Jun 2. PMID 19491241
- [Background] Turnbaugh PJ, Ley RE, Mahowald MA, Magrini V, Mardis ER, Gordon JI. An obesity-associated gut microbiome with increased capacity for energy harvest. Nature. 2006 Dec 21;444(7122):1027-31. doi: 10.1038/nature05414. PMID 17183312
- [Background] Sanchez M, Panahi S, Tremblay A. Childhood obesity: a role for gut microbiota? Int J Environ Res Public Health. 2014 Dec 23;12(1):162-75. doi: 10.3390/ijerph120100162. PMID 25546278
- [Background] Kadooka Y, Sato M, Imaizumi K, Ogawa A, Ikuyama K, Akai Y, Okano M, Kagoshima M, Tsuchida T. Regulation of abdominal adiposity by probiotics (Lactobacillus gasseri SBT2055) in adults with obese tendencies in a randomized controlled trial. Eur J Clin Nutr. 2010 Jun;64(6):636-43. doi: 10.1038/ejcn.2010.19. Epub 2010 Mar 10. PMID 20216555
- [Background] Chang BJ, Park SU, Jang YS, Ko SH, Joo NM, Kim SI, Kim CH, Chang DK. Effect of functional yogurt NY-YP901 in improving the trait of metabolic syndrome. Eur J Clin Nutr. 2011 Nov;65(11):1250-5. doi: 10.1038/ejcn.2011.115. Epub 2011 Jun 22. PMID 21697819
- [Background] Zarrati M, Salehi E, Nourijelyani K, Mofid V, Zadeh MJ, Najafi F, Ghaflati Z, Bidad K, Chamari M, Karimi M, Shidfar F. Effects of probiotic yogurt on fat distribution and gene expression of proinflammatory factors in peripheral blood mononuclear cells in overweight and obese people with or without weight-loss diet. J Am Coll Nutr. 2014;33(6):417-25. doi: 10.1080/07315724.2013.874937. Epub 2014 Jul 31. PMID 25079040
- [Background] Kang JH, Yun SI, Park HO. Effects of Lactobacillus gasseri BNR17 on body weight and adipose tissue mass in diet-induced overweight rats. J Microbiol. 2010 Oct;48(5):712-4. doi: 10.1007/s12275-010-0363-8. Epub 2010 Nov 3. PMID 21046354
- [Background] Piche T, des Varannes SB, Sacher-Huvelin S, Holst JJ, Cuber JC, Galmiche JP. Colonic fermentation influences lower esophageal sphincter function in gastroesophageal reflux disease. Gastroenterology. 2003 Apr;124(4):894-902. doi: 10.1053/gast.2003.50159. PMID 12671885
- [Background] Cani PD, Bibiloni R, Knauf C, Waget A, Neyrinck AM, Delzenne NM, Burcelin R. Changes in gut microbiota control metabolic endotoxemia-induced inflammation in high-fat diet-induced obesity and diabetes in mice. Diabetes. 2008 Jun;57(6):1470-81. doi: 10.2337/db07-1403. Epub 2008 Feb 27. PMID 18305141
- [Background] Cani PD, Delzenne NM. Interplay between obesity and associated metabolic disorders: new insights into the gut microbiota. Curr Opin Pharmacol. 2009 Dec;9(6):737-43. doi: 10.1016/j.coph.2009.06.016. Epub 2009 Jul 21. PMID 19628432
- [Background] Cani PD, Delzenne NM. The gut microbiome as therapeutic target. Pharmacol Ther. 2011 May;130(2):202-12. doi: 10.1016/j.pharmthera.2011.01.012. Epub 2011 Feb 2. PMID 21295072
- [Background] Pacifico L, Martino MD, Catalano C, Panebianco V, Bezzi M, Anania C, Chiesa C. T1-weighted dual-echo MRI for fat quantification in pediatric nonalcoholic fatty liver disease. World J Gastroenterol. 2011 Jul 7;17(25):3012-9. doi: 10.3748/wjg.v17.i25.3012. PMID 21799647
- [Background] Schwimmer JB, Middleton MS, Behling C, Newton KP, Awai HI, Paiz MN, Lam J, Hooker JC, Hamilton G, Fontanesi J, Sirlin CB. Magnetic resonance imaging and liver histology as biomarkers of hepatic steatosis in children with nonalcoholic fatty liver disease. Hepatology. 2015 Jun;61(6):1887-95. doi: 10.1002/hep.27666. Epub 2015 Feb 5. PMID 25529941
- [Background] Di Martino M, Pacifico L, Bezzi M, Di Miscio R, Sacconi B, Chiesa C, Catalano C. Comparison of magnetic resonance spectroscopy, proton density fat fraction and histological analysis in the quantification of liver steatosis in children and adolescents. World J Gastroenterol. 2016 Oct 21;22(39):8812-8819. doi: 10.3748/wjg.v22.i39.8812. PMID 27818597
- [Background] Szczepaniak LS, Nurenberg P, Leonard D, Browning JD, Reingold JS, Grundy S, Hobbs HH, Dobbins RL. Magnetic resonance spectroscopy to measure hepatic triglyceride content: prevalence of hepatic steatosis in the general population. Am J Physiol Endocrinol Metab. 2005 Feb;288(2):E462-8. doi: 10.1152/ajpendo.00064.2004. Epub 2004 Aug 31. PMID 15339742